CLINICAL TRIAL: NCT04092738
Title: ´Sit Less, Move More' at Work: Impact of a mHealth Intervention on the Glycaemic Control and Anthropometric Profile of Office Employees With Diabetes Type 2. A Randomized Controlled Trial.
Brief Title: ´Sit Less, Move More' at Work: mHealth Intervention on Office Employees With Diabetes Type 2.
Acronym: Walk@Work
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Consorci Hospitalari de Vic (Other); Institut Català de la Salut (Other); University of Vic - Central University of Catalonia (Other); Puerta de Hierro University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI17/01788
Record Dates: First submitted 2018-07-16; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type II
Keywords: mHealth; Physical Activity; Glucose, Blood; Glycated Hemoglobin A1c; Health-Related Quality Of Life; Quality of Life; Triglycerides; HDL Cholesterol; LDL Cholesterol; Blood Pressure, Arterial; Presenteeism; Sitting time; Sedentary Behaviour; Workplace
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention group, subjects will receive brief advice on occupational physical activity, sedentary behaviour and Diabetes Type 2. In addition, participants will be provided with an external movement sensor that will be linked to the Walk@WalkApp-Diab for Android and iOS. This App will monitor the time participants spend sitting, walking and standing during working hours. It will also provide participants with strategies to "sit less and move more" at work throughout 13 weeks. This mHealth intervention aims to change occupational sitting by replacing desk-based activities by active tasks.
  Interventions: Behavioral: Walk@WorkApp-Diab
- Control Group (No Intervention): Subjects will receive brief advice on occupational physical activity, sedentary behaviour and Diabetes Type 2.

INTERVENTIONS:
Behavioral: Walk@WorkApp-Diab — The intervention (Walk@WorkApp-Diab), based on an mHealth program, consists on replacing sedentary job tasks for active ones, during 13 weeks. The intervention group will download the mHealth program into their personal cellphones
  Other Names: mHealth intervention
  Arms: Intervention Group

SUMMARY:
The objective of the study is measuring the impact of a ´sit less, move more' mHealth intervention at work on the glycaemic control and anthropometric profile of office employees with diabetes type 2 (DT2) at short, mid and long term.

DETAILED DESCRIPTION:
A double-blind randomized controlled trial. Seven Primary Care Centers from Spain (n=5 Catalonia, n=2 Madrid), 2 hospitals (n=1 Catalonia, n=1 Madrid) and 2 companies (occupational health services; n=1 public, n=1 private) will participate in the study. In each center, physicians, nurses, endocrinologists and occupational physicians will recruit patients with DT2 who spend at least 55% of their working hours doing desk-based tasks (OSPAQ) and have a cellphone. Following the CONSORT Statement (2010), volunteers will be randomized into a control (CG) or intervention group (IG) by the research team using a computer program to generate the random sequence. 184 individuals are needed in each group. Main variables: fasting glucose levels, HbA1c, weight, height, BMI, waist circumference. Occupational sitting time and sitting time breaks will be measured using ActivPAL devices. Other variables: physical activity (IPAQ short), quality of life (EuroQool), presenteeism (WLQ), triglycerides, total cholesterol (LDL and HDL), blood pressure and sociodemographic variables.

Intervention: A mHealth program (13 wks) will progressively replace occupational sitting time with light physical activities. Participants from the CG will receive usual care. Multivariate analysis will assess changes over time (post intervention and at 6 months follow up) in the dependent variables; looking at differences between groups. Intention to treat will be applied.

ELIGIBILITY:
Inclusion Criteria:

* DM2 diagnosed office employees according to international criteria.
* Doing sedentary tasks during at least a 55% of their daily work schedule (according to the Occupational Sedentary and Physical Activity Questionnaire: OSPAQ >55%).
* Having a cellphone .
* Having a minimum work contract of 18.5 hours per week.
* Being able to get up from the chair or to walk by themselves (without any help).

Exclusion Criteria:

* Not having a cellphone.
* Having some pathology/disability/injury which changes their ability and capacity to walk or getting up from the chair.
* Doing less than a 55% of the daily tasks in a sitting position according to the OSPAQ questionnaire.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 368 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in Fasting glucose levels | Two measurement points: (a) Before the intervention starts, (b) at 6 months after intervention has finished
  Blood tests
Change in concentration of HbA1c | Two measurement points: (a) before the intervention starts, (b) at 6 months after intervention has finished.
  Blood tests
Change in weight | Three measurement points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after intervention has finished.
  Body weight in kilograms (electronic scale-Seca 899/217)
Change in height | Three measurement points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after intervention has finished.
  Body height in metres (electronic scale-Seca 899/217)
Change in Body Mass Index | Three measurement points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after intervention has finished.
  Weight and height will be combined to report Body Mass Index (kg/m2)
Change in Waist circumference | Three measurment points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after the intervention has finished
  Waist circumference in centimetres using a flexible steel tape (Seca 203)

SECONDARY OUTCOMES:
Change in objective Occupational sedentary behaviour | Three measurment points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after the intervention has finished.
  Total sitting time (minutes/day), sedendary bouts (daily time spent sitting on less than 20 minutes periods, between 20-60 minutes periods, more than 60 minutes period (ActivPal device)
Change in subjective domain-specific sedentary behaviour | Three measurment points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after the intervention has finished.
  Workforce Sitting Questionnaire (daily time spent sitting watching TV, working, at home, as transport and for leisure during working days and nonworking days (minutes/day)
Change in objective occupational physical activity | Three measurment points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after the intervention has finished.
  Minutes/day spent doing light and moderate-to-vigorous physical activity (ActivPal device)
Change in subjective occupational physical activity | Three measurment points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after the intervention has finished.
  Minutes/day walking, doing moderate and vigorous physical activity (International Physical Activity Questionnaire, IPAQ)

OTHER OUTCOMES:
Change in health-related quality of life | Three measurment points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after the intervention has finished.
  EQ-5d-3L. Scores range from 0 to 100 (0 describes the worse health you can imagine while 100 describes the best health you can imagine)
Change in Presenteeism levels | Three measurment points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after the intervention has finished.
  Work Limitations Questionnaire. Scores range from 0 to 100 (0 describes that your health dones not limit you at all in doing thw work tasks, while 100 describes your health limits you a lot your work tasks)
Change in concentration of Triglycerides | Two measurement points: (a) Before the intervention starts, (b) at 6 months after the intervention has finished.
  Blood tests (mg/dL)
Change in total cholesterol levels | Two measurement points: (a) Before the intervention starts, (b) at 6 months after the intervention has finished.
  Blood tests (mg/dL)
Change in blood pressure | Three measurment points: (a) before the intervention, (b) immediately after the intervention, (c) at 6 months after the intervention has finished.
  Digital automatic blood pressure monitor-Omron M7 (mmHg)
Sociodemographic variables (age, gender, socio economic status) | One measurment point: (a) before the intervention.
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anna Puig Ribera, Principal Investigator — Universitat de Vic; Carlos Martin Cantera, Study Chair — Jordi Gol i Gurina Foundation - IDIAP Jordi Gol; Francesc Alòs Colomer, Study Chair — Catalan Institute of Health; Mercè Solà Gonfaus, Study Chair — Catalan Institute of Health; Ana Urpí Fernández, Study Chair — Catalan Institute of Health; Josep Maria Molina Aragonés, Study Chair — Catalan Institute of Health; Blanca Funollet Santos, Study Chair — Catalan Institute of Health; Laura Illamola Martin, Study Chair — EAP Dreta de l'Eixample S.L.P; Ignasi Saigí Ullastre, Study Chair — Consorci Hospitalari de Vic (CHV); Emi Chirveches-Pérez, Study Chair — Consorci Hospitalari de Vic (CHV); Montserrat Martín-Horcajo, Study Chair — Universitat de Vic-Universitat Central de Catalunya (UVIC-UCC); Montserrat Munuera Grau, Study Chair — Catalan Institute of Health; Miguel Brito, Study Chair — Madrid Health Service; David Pérez Manchon, Study Chair — Madrid Health Service; María Lorena López Catañon, Study Chair — Madrid Health Service; Montserrat Solís Muñoz, Study Chair — Madrid Health Service; Judit Bort-Roig, Study Chair — University of Vic - Central University of Catalonia; Mireia Félez-Nóbrega, Study Chair — Parc Sanitari Sant Joan de Déu (Sant Boi de Llobregat); Francesc Garcia Cuyàs, Study Chair — Hospital Sant Joan de Déu (Barcelona)
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alos F, Colomer MA, Bort-Roig J, Martin-Cantera C, Minaya A, Saigi I, Sitjar-Suner M, Puig-Ribera A. Impact of a primary care-based mobile health intervention to 'sit less and move more' on HbA1c, blood pressure, and other clinical outcomes in office employees with type 2 diabetes: A randomized controlled trial. Prim Care Diabetes. 2025 Oct;19(5):434-445. doi: 10.1016/j.pcd.2025.05.010. Epub 2025 Jun 9. PMID 40494751
- [Derived] Alos F, Colomer MA, Martin-Cantera C, Solis-Munoz M, Bort-Roig J, Saigi I, Chirveches-Perez E, Sola-Gonfaus M, Molina-Aragones JM, Puig-Ribera A. Effectiveness of a healthcare-based mobile intervention on sedentary patterns, physical activity, mental well-being and clinical and productivity outcomes in office employees with type 2 diabetes: study protocol for a randomized controlled trial. BMC Public Health. 2022 Jun 29;22(1):1269. doi: 10.1186/s12889-022-13676-x. PMID 35768818
- [Derived] Bort-Roig J, Chirveches-Perez E, Garcia-Cuyas F, Dowd KP, Puig-Ribera A. Monitoring Occupational Sitting, Standing, and Stepping in Office Employees With the W@W-App and the MetaWearC Sensor: Validation Study. JMIR Mhealth Uhealth. 2020 Aug 4;8(8):e15338. doi: 10.2196/15338. PMID 32459625